CLINICAL TRIAL: NCT04881851
Title: Effects of Inositol Alone or Associated With Alpha-lipoic Acid in Polycystic Ovary Syndrome Treatment
Acronym: IALA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study treatment products expired
Sponsor: Universita di Verona (Other)
Collaborators: Laborest Italia SPA (Unknown)
Responsible Party: Principal Investigator, Paolo Moghetti, Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE10403
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Inositol; alpha-lipoic acid
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Inositol; Thioctic Acid; Folic Acid

STUDY DESIGN:
Intervention Model Description: Double blinded, three-armed RCT
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inositol + alpha lipoic acid (Experimental): Inositol 1000 mg + alpha lipoic acid 400 mg + folic acid 200 ug: 1 sachet at breakfast and 1 sachet at dinner
  Interventions: Dietary Supplement: Inositol + alpha lipoic acid
- Inositol (Experimental): Inositol 1000 mg + folic acid 200 ug: 1 sachet at breakfast and 1 sachet at dinner
  Interventions: Dietary Supplement: Inositol
- Folic acid (Placebo Comparator): Folic acid 200 ug: 1 sachet at breakfast and 1 sachet at dinner
  Interventions: Dietary Supplement: Folic acid (placebo comparator)

INTERVENTIONS:
Dietary Supplement: Inositol + alpha lipoic acid — Inositol 1000 mg + alpha lipoic acid 400 mg + folic acid 200 ug: 1 sachet at breakfast and 1 sachet at dinner
  Arms: Inositol + alpha lipoic acid
Dietary Supplement: Inositol — Inositol 1000 mg + folic acid 200 ug: 1 sachet at breakfast and 1 sachet at dinner
  Arms: Inositol
Dietary Supplement: Folic acid (placebo comparator) — Folic acid 200 ug: 1 sachet at breakfast and 1 sachet at dinner
  Arms: Folic acid

SUMMARY:
The aim of this double-blinded, three-armed randomized controlled trial (RCT) is to evaluate the effects of a 6 months treatment with inositol alone or inositol associated with alpha-lipoic acid in women with polycystic ovary syndrome (PCOS).

The study population is composed of 90 women with PCOS (diagnosed according to the Rotterdam criteria). Subjects are randomized to one of the 3 arms of treatment (Inositol + alpha lipoic acid + folic acid vs inositol + folic acid vs folic acid alone).

At recruitment and after 6 months of treatment, the following data are collected:

* clinical data: height, weight, BMI, waist and hip circumference, blood pressure, Ferriman Gallwey Score, menstrual diary
* endocrine parameters (serum total and free testosterone levels, SHBG levels)
* metabolic profile: glycemia and insulinemia at fasting and after oral glucose tolerance test (OGTT), serum lipids
* insulin-sensitivity measured by the hyperinsulinemic-euglycemic clamp and surrogate indexes
* ovarian ultrasound data. Furthermore, ovulation is evaluated from the 2nd to the 6th month of the study through progesterone serial dosages on weekly urinary samples.

The primary outcome of the study is the serum free testosterone variation after 6 months of treatment. Secondary outcomes are the variations of lipid profile, ovarian morphology and insulin-sensitivity after 6 months and the number of ovulations occurring in the last 4 months of treatment.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effects of a 6 months treatment with inositol, alone or associated with alpha-lipoic acid, in women with PCOS. This is a double blinded, three-armed RCT.

The study population is composed of 90 women with PCOS, recruited at the Department of Endocrinology and Metabolic Disease of Azienda Ospedaliera Universitaria Integrata (AOUI), Verona.

After recruitment, subjects are randomly assigned to one of the 3 arms of treatment (Inositol + alpha lipoic acid + folic acid vs inositol + folic acid vs folic acid alone). Randomisation is stratified by BMI category (3 categories 18<BMI<25, 25≥BMI<30, 30≥BMI<35 Kg/m2); randomisation list is generated by the statistical software Stata 13.1.

At baseline and after 6 months of treatment, the following data are collected:

* clinical examination: family and personal medical history, menstrual diary, physical examination including height, weight, waist and hip circumferences, blood pressure and hirsutism score (modified Ferriman-Gallwey score)
* total and free testosterone and sex hormone binding globulin (SHBG) blood levels, evaluated in the early follicular phase or after 3 months of amenorrhea
* metabolic profile: glycemia and insulinemia at fasting and after 2h OGTT, serum lipids (total cholesterol, HDL-cholesterol and triglycerides). Glycemia and insulinemia values during OGTT will be used to calculate surrogate indexes of insulin resistance
* insulin-sensitivity measured by the hyperinsulinemic-euglycemic clamp technique. Data obtained with this test will be normalized for lean mass, measured by bioelectrical impedance. The hyperinsulinemic-euglycemic clamp is repeated after 6 months of treatment only in subjects who are insulin-resistant at baseline (M-value < 8.6 mg/kg min).
* Chronic inflammation markers (CRP)
* Ovarian ultrasound evaluation, including measurement of the 3 diameters for ovarian volume calculation, and follicle count. The ultrasound examination will be executed by a gynaecologist at the Department of Gynaecology and Obstetrics at AOUI, Verona.

Furthermore, all the study participants are subjected to:

* ovulation assessment by serial progesterone dosages on weekly urinary samples. Patients are given numbered urine beakers and are instructed to collect night urine weekly, starting at the 3rd month of treatment and until the end of the study (17 samples).
* monitoring visits after 2 and 4 months of treatment, to evaluate therapy compliance and possible adverse events.

  30 ml blood samples of the study participants will be preserved for 10 years. On these samples, further examinations will be considered if new important markers of PCOS will emerge in the future.

ELIGIBILITY:
Inclusion Criteria:

* female subjects
* age between 18 and 40 years old
* diagnosed with PCOS (according to the Rotterdam criteria)
* not use of possible interfering drugs in the 4 previous months
* written informed consent.

Exclusion Criteria:

* BMI ≥ 35 kg/m2
* acute illnesses
* chronic kidney or hepatic disease
* pregnant
* taking possible interfering drugs

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Free testosterone variation | 6 months
  Free testosterone variation after 6 months of treatment

SECONDARY OUTCOMES:
Insulin sensitivity variation | 6 months
  Insulin sensitivity variation after 6 months of treatment, evaluated by surrogate indexes in all the subjects and by repeating hyperinsulinemic euglycemic clamp after 6 months of treatment in women that are insulin-resistant at baseline
Lipid profile variation | 6 months
  Lipid profile variation after 6 months of treatment
Ovarian morphology variation | 6 months
  Ovarian morphology variation after 6 months of treatment
Number of ovulations in the last 4 months of treatment | 4 months
  Number of ovulations in the last 4 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Moghetti, Professor, Principal Investigator — Università degli studi di Verona
Locations (1):
- Endocrinology, Diabetes and Metabolism Section, Department of Medicine, University of Verona and Azienda Ospedaliera Universitaria Integrata of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in publications will be shared
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available when the study will be completed. They will remain available for 3 years.
Access Criteria: Upon specified request.

REFERENCES:
- [Background] Franks S. Polycystic ovary syndrome. N Engl J Med. 1995 Sep 28;333(13):853-61. doi: 10.1056/NEJM199509283331307. No abstract available. PMID 7651477
- [Background] Dunaif A. Insulin resistance and the polycystic ovary syndrome: mechanism and implications for pathogenesis. Endocr Rev. 1997 Dec;18(6):774-800. doi: 10.1210/edrv.18.6.0318. PMID 9408743
- [Background] Baptiste CG, Battista MC, Trottier A, Baillargeon JP. Insulin and hyperandrogenism in women with polycystic ovary syndrome. J Steroid Biochem Mol Biol. 2010 Oct;122(1-3):42-52. doi: 10.1016/j.jsbmb.2009.12.010. Epub 2009 Dec 28. PMID 20036327
- [Background] De Leo V, la Marca A, Petraglia F. Insulin-lowering agents in the management of polycystic ovary syndrome. Endocr Rev. 2003 Oct;24(5):633-67. doi: 10.1210/er.2002-0015. PMID 14570747
- [Background] Nestler JE, Jakubowicz DJ, Evans WS, Pasquali R. Effects of metformin on spontaneous and clomiphene-induced ovulation in the polycystic ovary syndrome. N Engl J Med. 1998 Jun 25;338(26):1876-80. doi: 10.1056/NEJM199806253382603. PMID 9637806
- [Background] Moghetti P, Castello R, Negri C, Tosi F, Perrone F, Caputo M, Zanolin E, Muggeo M. Metformin effects on clinical features, endocrine and metabolic profiles, and insulin sensitivity in polycystic ovary syndrome: a randomized, double-blind, placebo-controlled 6-month trial, followed by open, long-term clinical evaluation. J Clin Endocrinol Metab. 2000 Jan;85(1):139-46. doi: 10.1210/jcem.85.1.6293. PMID 10634377
- [Background] Fleming R, Hopkinson ZE, Wallace AM, Greer IA, Sattar N. Ovarian function and metabolic factors in women with oligomenorrhea treated with metformin in a randomized double blind placebo-controlled trial. J Clin Endocrinol Metab. 2002 Feb;87(2):569-74. doi: 10.1210/jcem.87.2.8261. PMID 11836287
- [Background] Azziz R, Ehrmann D, Legro RS, Whitcomb RW, Hanley R, Fereshetian AG, O'Keefe M, Ghazzi MN; PCOS/Troglitazone Study Group. Troglitazone improves ovulation and hirsutism in the polycystic ovary syndrome: a multicenter, double blind, placebo-controlled trial. J Clin Endocrinol Metab. 2001 Apr;86(4):1626-32. doi: 10.1210/jcem.86.4.7375. PMID 11297595
- [Background] Tang T, Lord JM, Norman RJ, Yasmin E, Balen AH. Insulin-sensitising drugs (metformin, rosiglitazone, pioglitazone, D-chiro-inositol) for women with polycystic ovary syndrome, oligo amenorrhoea and subfertility. Cochrane Database Syst Rev. 2012 May 16;(5):CD003053. doi: 10.1002/14651858.CD003053.pub5. PMID 22592687
- [Background] Thessaloniki ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Consensus on infertility treatment related to polycystic ovary syndrome. Hum Reprod. 2008 Mar;23(3):462-77. doi: 10.1093/humrep/dem426. PMID 18308833
- [Background] Barua S, Kuizon S, Junaid MA. Folic acid supplementation in pregnancy and implications in health and disease. J Biomed Sci. 2014 Aug 19;21(1):77. doi: 10.1186/s12929-014-0077-z. PMID 25135350
- [Background] Saltiel AR. Second messengers of insulin action. Diabetes Care. 1990 Mar;13(3):244-56. doi: 10.2337/diacare.13.3.244. PMID 2137771
- [Background] Baillargeon JP, Diamanti-Kandarakis E, Ostlund RE Jr, Apridonidze T, Iuorno MJ, Nestler JE. Altered D-chiro-inositol urinary clearance in women with polycystic ovary syndrome. Diabetes Care. 2006 Feb;29(2):300-5. doi: 10.2337/diacare.29.02.06.dc05-1070. PMID 16443877
- [Background] Fenkci V, Fenkci S, Yilmazer M, Serteser M. Decreased total antioxidant status and increased oxidative stress in women with polycystic ovary syndrome may contribute to the risk of cardiovascular disease. Fertil Steril. 2003 Jul;80(1):123-7. doi: 10.1016/s0015-0282(03)00571-5. PMID 12849813
- [Background] Giordano D, Corrado F, Santamaria A, Quattrone S, Pintaudi B, Di Benedetto A, D'Anna R. Effects of myo-inositol supplementation in postmenopausal women with metabolic syndrome: a perspective, randomized, placebo-controlled study. Menopause. 2011 Jan;18(1):102-4. doi: 10.1097/gme.0b013e3181e8e1b1. PMID 20811299
- [Background] Capasso I, Esposito E, Maurea N, Montella M, Crispo A, De Laurentiis M, D'Aiuto M, Frasci G, Botti G, Grimaldi M, Cavalcanti E, Esposito G, Fucito A, Brillante G, D'Aiuto G, Ciliberto G. Combination of inositol and alpha lipoic acid in metabolic syndrome-affected women: a randomized placebo-controlled trial. Trials. 2013 Aug 28;14:273. doi: 10.1186/1745-6215-14-273. PMID 23981814
- [Background] Jacob S, Ruus P, Hermann R, Tritschler HJ, Maerker E, Renn W, Augustin HJ, Dietze GJ, Rett K. Oral administration of RAC-alpha-lipoic acid modulates insulin sensitivity in patients with type-2 diabetes mellitus: a placebo-controlled pilot trial. Free Radic Biol Med. 1999 Aug;27(3-4):309-14. doi: 10.1016/s0891-5849(99)00089-1. PMID 10468203
- [Background] Nestler JE, Jakubowicz DJ, Reamer P, Gunn RD, Allan G. Ovulatory and metabolic effects of D-chiro-inositol in the polycystic ovary syndrome. N Engl J Med. 1999 Apr 29;340(17):1314-20. doi: 10.1056/NEJM199904293401703. PMID 10219066
- [Background] Iuorno MJ, Jakubowicz DJ, Baillargeon JP, Dillon P, Gunn RD, Allan G, Nestler JE. Effects of d-chiro-inositol in lean women with the polycystic ovary syndrome. Endocr Pract. 2002 Nov-Dec;8(6):417-23. doi: 10.4158/EP.8.6.417. PMID 15251831
- [Background] Gerli S, Mignosa M, Di Renzo GC. Effects of inositol on ovarian function and metabolic factors in women with PCOS: a randomized double blind placebo-controlled trial. Eur Rev Med Pharmacol Sci. 2003 Nov-Dec;7(6):151-9. PMID 15206484
- [Background] Cheang KI, Baillargeon JP, Essah PA, Ostlund RE Jr, Apridonize T, Islam L, Nestler JE. Insulin-stimulated release of D-chiro-inositol-containing inositolphosphoglycan mediator correlates with insulin sensitivity in women with polycystic ovary syndrome. Metabolism. 2008 Oct;57(10):1390-7. doi: 10.1016/j.metabol.2008.05.008. PMID 18803944
- [Background] Masharani U, Gjerde C, Evans JL, Youngren JF, Goldfine ID. Effects of controlled-release alpha lipoic acid in lean, nondiabetic patients with polycystic ovary syndrome. J Diabetes Sci Technol. 2010 Mar 1;4(2):359-64. doi: 10.1177/193229681000400218. PMID 20307398
- [Background] Elnashar A, Abdelmageed E, Fayed M, Sharaf M. Clomiphene citrate and dexamethazone in treatment of clomiphene citrate-resistant polycystic ovary syndrome: a prospective placebo-controlled study. Hum Reprod. 2006 Jul;21(7):1805-8. doi: 10.1093/humrep/del053. Epub 2006 Mar 16. PMID 16543255
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Background] Kozakowski J, Zgliczynski W. Body composition, glucose metabolism markers and serum androgens - association in women with polycystic ovary syndrome. Endokrynol Pol. 2013;64(2):94-100. PMID 23653271
- [Background] Hatch R, Rosenfield RL, Kim MH, Tredway D. Hirsutism: implications, etiology, and management. Am J Obstet Gynecol. 1981 Aug 1;140(7):815-30. doi: 10.1016/0002-9378(81)90746-8. PMID 7258262
- [Background] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510
- [Background] Moghetti P, Tosi F, Castello R, Magnani CM, Negri C, Brun E, Furlani L, Caputo M, Muggeo M. The insulin resistance in women with hyperandrogenism is partially reversed by antiandrogen treatment: evidence that androgens impair insulin action in women. J Clin Endocrinol Metab. 1996 Mar;81(3):952-60. doi: 10.1210/jcem.81.3.8772557.
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] Gray DS, Bray GA, Gemayel N, Kaplan K. Effect of obesity on bioelectrical impedance. Am J Clin Nutr. 1989 Aug;50(2):255-60. doi: 10.1093/ajcn/50.2.255. PMID 2756912
- [Background] Carlomagno G, Unfer V. Inositol safety: clinical evidences. Eur Rev Med Pharmacol Sci. 2011 Aug;15(8):931-6. PMID 21845803
- [Background] Shay KP, Moreau RF, Smith EJ, Smith AR, Hagen TM. Alpha-lipoic acid as a dietary supplement: molecular mechanisms and therapeutic potential. Biochim Biophys Acta. 2009 Oct;1790(10):1149-60. doi: 10.1016/j.bbagen.2009.07.026. Epub 2009 Aug 4. PMID 19664690
- [Background] Bae SM, Bae MN, Kim EY, Kim IK, Seo MW, Shin JK, Cho SR, Jeong GH. Recurrent Insulin Autoimmune Syndrome Caused by alpha-Lipoic Acid in Type 2 Diabetes. Endocrinol Metab (Seoul). 2013 Dec;28(4):326-30. doi: 10.3803/EnM.2013.28.4.326. Epub 2013 Dec 12. PMID 24396698